CLINICAL TRIAL: NCT04809051
Title: Don't Throw Your Heart Away: Patient Study 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Gretchen Chapman, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1 F30 HL152526-01-D; 1F30HL152526-01 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Transplant Disorder
Keywords: Heart Transplant; Transplant Survival; Applied Ethics; Medical Student; Human Behavior; Decision Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1: Combined Transplant Pictograph (No Intervention): Participants randomized to baseline (control) arm Condition 1 will view only combined transplant survival outcome information (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center) when making a choice between the two hospitals. The "survival following transplant" metric is displayed as a survival rate pictograph corresponding to all patients at the center who received transplants.
- Condition 2: Stratified Transplant Pictograph (Experimental): Participants randomized to Condition 2 will view only stratified transplant survival outcome information when making a choice between the two hospitals. The "survival following transplant" metric is displayed as a pair of survival rate pictographs corresponding to two distinct groups of transplant patients at the center: those who received optimal donor organs and those who received adequate donor organs.
  Interventions: Other: Stratified Transplant Survival Metric
- Condition 3: Combined Transplant SRTR (Experimental): Participants randomized to Condition 3 will view only combined transplant survival outcome information (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center) when making a choice between the two hospitals. The "survival following transplant" metric is displayed as a quintile score corresponding to all patients at the center who received transplants.
  Interventions: Other: SRTR Information Format
- Condition 4: Stratified Transplant SRTR (Experimental): Participants randomized to Condition 4 will view only stratified transplant survival outcome information when making a choice between the two hospitals. The "survival following transplant" metric is displayed as a pair of quintile scores corresponding to two distinct groups of transplant patients at the center: those who received optimal donor organs and those who received adequate donor organs.
  Interventions: Other: Stratified Transplant Survival Metric; Other: SRTR Information Format

INTERVENTIONS:
Other: Stratified Transplant Survival Metric — Both transplant metric conditions display the number of hearts offered to each center, the number of hearts accepted by each center, and the number of transplants performed at each center (in a year), in addition to the condition-specific metrics below. The stratified condition instead features a pair of values corresponding to each center's offers/acceptances/transplant survival rates for donor hearts of "optimal" or "adequate" quality.
  Arms: Condition 2: Stratified Transplant Pictograph; Condition 4: Stratified Transplant SRTR
Other: SRTR Information Format — The information format varies based on how the transplant hospital statistics are organized when presented to participants on the choice screen. The SRTR conditions mimic the information format present on the SRTR public reporting website.
  Arms: Condition 3: Combined Transplant SRTR; Condition 4: Stratified Transplant SRTR

SUMMARY:
This empirical study tests whether transplant center performance data that reflect center donor acceptance rates influence patients and their family members to evaluate centers with high organ decline rates less favorably than centers with low organ decline rates. 400 transplant patients and family members will be recruited from transplant support group social media websites and randomized to one of four different information presentation conditions. Upon viewing a pair of outcome tables corresponding to their condition, the participants are asked to choose which hospital is higher performing (one hospital with a non-selective "accepting" strategy and one hospital with a more selective "cherrypicking" strategy.

ELIGIBILITY:
Inclusion Criteria:

Participants will be asked to participate if they confirm the following inclusion criteria in the consent form.

1. 18 years of age or older
2. must read and understand the information in the consent form
3. must want to participate in the research and continue with the survey
4. must be a pre- or post-transplant patient or family member of the transplant patient

Exclusion Criteria:

Participants who do not meet the primary criterion of being a pre- or post-transplant patient or family member of the transplant patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Hospital Choice | 1 day
  The outcome variable will be a measure of binary choice between two hospitals: one with a selective donor-heart acceptance strategy and one with a non-selective donor heart acceptance strategy.
  Participants will respond to the question "Which Hospital is higher performing? Please click on one of the two tables below to indicate which hospital is the better choice." Participants will choose been two outcome tables featuring the selective and non-selective hospital (counterbalanced, such that each of the two choices is equally likely to be presented at top of the choice scenario in each condition). The number of participants that choose each hospital will be the measured outcome variable used in analyses.

SECONDARY OUTCOMES:
Mediator of Hospital Choice | 1 day
  On the next page of the survey, participants will respond to three mediator questions: "There are many reasons why one transplant hospital might outperform another. Which reasons were most important in your decision? Please move the slider to indicate how much you considered each of the reasons below (0=reason was not important, 100=reason was extremely important)."
  Participants will then move a slider bar (0-100) to indicate the importance of the following three items:
  Patients were more likely to receive an excellent donor heart at the hospital I picked.
  Patients were less likely to receive a marginal donor heart at the hospital I picked.
  Patients were more likely to receive any kind of heart at the hospital I picked.
  The third item (more likely to receive any kind of heart) will be the only variable that is included in the planned mediation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Butler, MS, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes The PI will make all of the raw IPD files - together with statistical analysis protocol descriptions and information for proper analysis available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts. All human subjects data are anonymized immediately when they are initially written from the online survey platform to the server, and thus participant confidentiality will not be compromised by this plan for data sharing.
  All hypotheses, methods, and planned analyses for the applicant's studies will be pre-registered on ClinicalTrials.gov and Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All of the raw files, statistical analysis protocol descriptions, and information for proper analysis will be available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts.
URL: https://osf.io/weqvj/